CLINICAL TRIAL: NCT05890053
Title: A 52-week, Open Phase III Study Evaluating the Long-term Safety and Efficacy of HSK16149 Capsules in Chinese Patients With Peripheral Neuralgia
Brief Title: To Evaluate the Long-term Safety and Efficacy of HSK16149 in Chinese Patients With Peripheral Neuralgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSK16149-303
Record Dates: First submitted 2023-02-26; First posted 2023-06-06 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2023-04

CONDITIONS: Peripheral Neuropathic Pain
MeSH Terms: interventions — BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HSK16149 40mg BID (Experimental): HSK16149 40mg , orally twice a day, treatment period; 52-weeks fixed dose.
  Interventions: Drug: HSK16149 40mg BID

INTERVENTIONS:
Drug: HSK16149 40mg BID — HSK16149 40mg ， orally twice a day, treatment period; 52-weeks fixed dose.
  Other Names: HSK16149

SUMMARY:
Investigate the long-term(52 weeks) safety and efficacy of HSK16149 capsules in Chinese patients with periphcral neuralgia

DETAILED DESCRIPTION:
Investigate the long-term(52 weeks) safety and efficacy of HSK16149 capsules in Chinese patients with Peripheral neuropathic pain

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who completed double-blind treatment and safety follow-up in HSK16149-201/301.
2. Able to understand and voluntarily sign informed consent.

Exclusion Criteria:

1. Medication compliance was < 80% in double-blind studies.
2. In double-blind study, EOT visit (V10) eGFR< 60 mL/min//1.73m2
3. Significant safety concerns or adverse events that did not recover before taking the drug in this study arose in the double-blind study.
4. Hepatitis B Surface antigen (HBsAg) positive or hepatitis C virus antibody (HCV Ab) positive during screening [further hepatitis B virus deoxyribonucleic acid (HBV DNA) titer detection or hepatitis C virus ribonucleic acid (HCV RNA) detection (beyond the detection limit of assay need to be excluded)], human immunodeficiency virus antibody (HIV) Ab) positive, serum antibody to treponema pallidum (TP Ab) positive (further test for treponema pallidum titer, if positive, excluded).
5. Women who are pregnant, planning to become pregnant during the study, or breastfeeding; Participants were not expected to use reliable contraceptive methods (including condoms, spermicides, or intrauterine devices) for 28 days after signing up for the ICF or planning to use progester-containing contraceptives during this period.
6. The researcher judged that the study could not be completed according to the scheme or that it was difficult to participate in the study due to safety.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the long-term safety of HSK16149 capsules in Chinese patients with peripheral neuralgia. | From week 1 to week 53
  Safety assessment variables included AE, ECG, laboratory test values, height and weight, physical examination, and vital signs. Safety data will be summarized by aggregate in SS and all subjects will be listed. Overall description of all AE occurred in subjects by total, and summary of cases, cases and percentage. Clinical judgments of laboratory indicators before and after drug administration (according to the range of normal values or the investigator's judgment of clinical significance) were summarized in the form of crosstabs, and the number and percentage of cases were calculated.

SECONDARY OUTCOMES:
Changes in SF-MPQ scores from baseline before and after treatment to evaluate the long-term effectiveness of HSK16149. | From week 1 to week 53
  Based on FAS, descriptive statistical analysis and mapping analysis were performed on the mean values of VAS, PRI and PPI scores and the mean changes from baseline of each visiting point, to compare whether there were statistical differences before and after treatment. Participants rate their pain in three parts of the questionnaire, which are combined into a single pain intensity score:
  Part 1 - fifteen descriptors of pain intensity, on a scale of 0 (none) to 3 (severe) Part 2 - a visual analog scale (VAS), in which the participant rates pain on a 100 mm-long horizontal line, where 0 mm = no pain and 100 mm = worst possible pain Part 3 - a Present Pain Intensity index in which the participant rates present pain intensity on a scale of 0 (no pain) to 5 (most intense pain)

CONTACTS AND LOCATIONS:
Locations (24):
- China (24):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Pinggu District Hospital, Beijing, Beijing Municipality
  - Emergency General Hospital, Beijing, Beijing Municipality
  - The Three Gorges Hospital Affiliated to Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Cangzhou People's Hospital, Cangzhou, Hebei
  - The Third Hospital of Hebei Medical University, Shijiangzhuang, Hebei
  - Kaifeng Hospital of Traditional Chinese Medicine, Kaifeng, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Nanyang First People's Hospital, Nanyang, Henan
  - Wuhan Central Hospital, Wuhan, Hubei
  - Nanjing First People's Hospital, Nanjing, Jiangsu
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Baotou Central Hospital, Baotou, Neimenggu
  - Jinan Central Hospital, Jinan, Shandong
  - The First Affiliated Hospital of Xi'an Medical University, Xi’an, Shanxi
  - Yuncheng Central Hospital, Yuncheng, Shanxi
  - The Second People's Hospital of Yibin, Yibin, Sichuan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Taizhou First People's Hospital, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No